CLINICAL TRIAL: NCT00952952
Title: A Randomized, Dose Ranging Trial of Mesalmine for the Treatment of Active Microscopic Colitis.
Brief Title: Trial of Mesalamine for the Treatment of Active Microscopic Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Paul E. Evans MD (Unknown); William J. Sandborn MD (Unknown); Edward V. Loftus MD (Unknown); Thomas C. Smryk MD (Unknown); Willaim Tremaine MD (Unknown)
Responsible Party: Darrell S. Pardi MD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-003637; evans 06
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Microscopic Colitis; Diarrhea
MeSH Terms: conditions — Colitis, Microscopic; Diarrhea | interventions — Mesalamine

INTERVENTIONS:
Drug: Mesalamine

SUMMARY:
Subjects must be 18 years old and older, have diarrhea and microscopic colitis. Pregnant or nursing females are excluded. They can't have other untreated diarrheal conditions. Subjects will receive medication for 8 weeks, followed by sigmoidoscopy with biopsies. The subjects will be monitored weekly. A pathologist will review pre and post treatment biopsies. Subjects that show improvement will be followed for 4 weeks post medication.

DETAILED DESCRIPTION:
We propose a prospective, randomized trial of mesalamine at 1.2g and 4.8g doses for the treatment of microscopic colitis. Our hypothesis is mesalamine is safe and effective for the treatment of diarrhea in microscopic colitis and that the 4.8g dose is more effective than the 1.2g dose.

We will recruit 70 subjects. The subjects will be randomized into to two groups, 4.8g dose, and 1.2g dose groups. Subjects will receive medication for 8 weeks, followed by sigmoidoscopy with biopsies. The subjects will be monitored weekly. A pathologist will review pre and post treatment biopsies. Responders will be followed for 4 weeks post medication.

Subjects must be 18 years old and older, have diarrhea and microscopic colitis. Subjects will be excluded if they have unsuccessful treatment or side effects to 5-ASA drugs, oral corticosteroids, or salicylate. and antibiotics, mesalamine, bismuth or steroid use in the last two weeks. Subjects may not be on anticholinergics, cholestyramine, digoxin. Pregnant or nursing females are excluded. They can't have other untreated diarrheal conditions.

A two-sample z-score test for proportions will be used to test whether relief rates are different between groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years old and older.
* Have diarrhea and microscopic colitis.
* They need to have a colon biopsy done at the Mayo Clinic in Rochester, MN within a year of enrollment.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of mesalamine at 1.2g and 4.8g doses in microscopic colitis for providing relief of diarrhea

SECONDARY OUTCOMES:
To compare the safety and tolerability of mesalamine at 1.2g and 4.8g doses in patients with microscopic colitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States